CLINICAL TRIAL: NCT03025204
Title: Enamel Matrix Proteins in the Treatment of Intrabony Defects in Patients With Aggressive and Chronic Periodontitis: Randomized Clinical Trial
Brief Title: Enamel Matrix Proteins in the Treatment of Intrabony Defects in Patients With Aggressive and Chronic Periodontitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Enilson Antonio Sallum, Professor Enilson Antonio Sallum, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 118/2015
Record Dates: First submitted 2017-01-16; First posted 2017-01-19 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2017-01

CONDITIONS: Aggressive Periodontitis
Keywords: Regeneration Procedures; Intrabony Defects; Cronic Periodontitis
MeSH Terms: conditions — Aggressive Periodontitis | interventions — enamel matrix proteins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- GAP Surgical Access (GAP + OFD, 15 patients) (Active Comparator): Patients diagnosed with generalized aggressive periodontitis (GAP), in which the previously selected intrabony defect will receive will receive open flap debridement.
  Interventions: Procedure: Open Flap Debridement
- GAP Surgical Access + EMD (GAP + OFD/EMD, 15 patients) (Experimental): Patients with a diagnosis of generalized aggressive periodontitis (GAP), in which the previously selected intrabony defect will receive open flap debridement and, in addition, application of the EMD in the defect.
  Interventions: Biological: Enamel Matrix Proteins; Procedure: Open Flap Debridement
- GCP Surgical Access + EMD (GCP + OFD/EMD, 15 patients) (Active Comparator): Patients with a diagnosis of generalized chronic periodontitis (GCP), in which the previously selected intrabony defect will receive open flap debridement and, in addition, application of the EMD in the defect.
  Interventions: Biological: Enamel Matrix Proteins; Procedure: Open Flap Debridement

INTERVENTIONS:
Biological: Enamel Matrix Proteins — EMD is composed of different proteins, 90% of which are amelogenins, which has the capacity to induce processes involved in the regeneration of periodontal tissues in a manner similar to normal tissue development (48). Several clinical and animal model studies have demonstrated the use of enamel matrix-derived proteins in regenerative periodontal procedures for the formation of a new periodontium.
  Arms: GAP Surgical Access + EMD (GAP + OFD/EMD, 15 patients); GCP Surgical Access + EMD (GCP + OFD/EMD, 15 patients)
Procedure: Open Flap Debridement — After administration of local anesthetics, full-thickness flaps will be raised in order to access all defect faces. Sulcular incisions will be performed extending to mesial and distal adjacent teeth, including the entire papilla in the flap. No relaxing incisions will be performed. All granulation tissue will then be carefully removed, and subsequently scaling and root planing will be performed. The surgical area will be irrigated with 0.9% saline and carefully inspected to ensure that all steps have been satisfactorily performed until then.

SUMMARY:
Approaches and objectives related to the treatment of patients with aggressive periodontitis are not markedly different compared patients with the chronic form. However, the large bone loss related to young age in this aggressive form, justify a well-founded strategy, intending to further stabilization of disease progression. For this, should make use of regenerative therapies in the advanced stages of treatment. Noteworthy is the use of proteins derived from the enamel matrix (EMD) in patients with chronic periodontitis, but there is little evidence about the effects of this material in aggressive periodontitis. Thus, the present study aims to evaluate the use of EMD in patients with aggressive periodontitis, comparing them to individuals with chronic periodontitis. Will then be selected 45 subjects, among patients with generalized chronic periodontitis (GCP) and generalized aggressive periodontitis (GAP), with one or more intra-bony defects in radiographic examination, with a minimum size of 4 mm deep and 2 mm horizontal, associated with a probing depth (PD) ≥6mm, to be treated according to the groups: GAP+OFD (n = 15) GAP patients which will receive open flap debridement; GAP+OFD/EMD (n=15) GAP patients which will receive open flap debridement and application of EMD; GCP+OFD/EMD (n=15) GCP patients which will receive open flap debridement and application of EMD. Clinical evaluations will be performed at baseline, 3, 6 months and 1 year after. At baseline, 7, 15, 45 days, 3, 6 months and 1 year after will be collect samples of gingival fluid to detect bone markers by Luminex / MAGpix technology. For the periods baseline, 3, 6 months and 1 year will be collected subgingival biofilm for the detection and quantification of periodontal pathogens by real-PCR. Will still be carried x-rays on baseline, 6 months and 1 year after, and questionnaires about patient satisfaction and perception of therapy at baseline, 7 days and 6 months. To compare the parameters evaluated, ANOVA, Tukey, chi-square, Spearman and Person tests will be used (α = 5%).

DETAILED DESCRIPTION:
General work plan and experimental methodology

1. Sample Selection

   After submission and approval of this project to the Research Ethics Committee (CEP) of the Piracicaba Dental School - UNICAMP, will be selected among the patients who seek spontaneously treatment in clinics pos graduate FOP-UNICAMP (where also will be performed the clinical phase of the study), 45 patients according to the inclusion criteria
2. Sampling Calculus

   The sample size required for each group was calculated considering the clinical attachment level (CAL) as the primary variable. To detect a difference of 1 mm with 5% alpha between groups, considering a standard deviation of 1 mm error and 80% test power, at least 12 patients in each group will be required. Considering that some patients may be lost during follow-up, 15 patients will be included in the present study.
3. Randomization and Blinding

   The examiner will be blind to the treatments. This is achieved by determining that the assessments are made by a professional not involved in the treatment. The division of patients into a group should be done by lot to be an entirely random sample, with treatments being randomly distributed among patients. Brown envelopes will be used, at the time of the surgical procedure, containing information from the treatment group that was generated through a computerized system.
4. Study design

   A parallel study will be carried out on 45 patients, with a duration of one year. The patients selected will be divided into 3 groups, whose teeth will receive the proposed treatments, as follows:
   * Group GAP Surgical Access (GAP + OFD, 15 patients) - Patients diagnosed with generalized aggressive periodontitis (PAG), in which the previously selected intrabony defect will receive will receive open flap debridement.
   * Group GAP Surgical Access + EMD (GAP + OFD/EMD, 15 patients) - Patients with a diagnosis of generalized aggressive periodontitis (PAG), in which the previously selected intrabony defect will receive open flap debridement and, in addition, application of the EMD in the defect.
   * Group GCP Surgical Access + EMD (GCP + OFD/EMD, 15 patients) - Patients with a diagnosis of generalized chronic periodontitis (PCG), in which the previously selected intrabony defect will receive open flap debridement and, in addition, application of the EMD in the defect.
5. Pre-surgical phase

   Initial examination: Selection of patients according to pre-established criteria.

   Initial Therapy: All patients will be educated about the causes and consequences of periodontal disease as well as on preventive techniques, including technique of sulcular brushing and flossing. Individuals will be given soft brushes in conjunction with a fluoride toothpaste, which will be replenished as needed. Professional removal of biofilm and supragingival calculus will be performed, as well as biofilm retention factors, if necessary.

   Treatment: Scaling anda root planing of all the teeth that present an indication. After the active phase of the treatment, patients will be included in supportive therapy with biweekly controls in the first month and monthly, until the end of the study, containing hygiene orientation, prophylaxis and quarterly retreatment of teeth that have a depth of probing greater than 5 mm, with BoP.
6. Surgical phase

   Teeth that present residual probing depth ≥ 6mm associated with radiographic evidence of intraboby deffects, according to the inclusion criteria mentioned above, will be included in the surgical procedure. Regenerative procedures will only be scheduled when all necessary non-surgical procedures are performed in concomitance with adequate PI and GI levels of up to 20%. All surgical procedures will be performed by the same operator. One hour before therapy, patients will receive a single dose of dexamethasone 4mg.

   Description of the technique: After administration of local anesthetics, full-thickness flaps will be raised in order to access all defect faces. Sulcular incisions will be performed extending to mesial and distal adjacent teeth, including the entire papilla in the flap. No relaxing incisions will be performed. All granulation tissue will then be carefully removed, and subsequently scaling and root planing will be performed. The surgical area will be irrigated with 0.9% saline and carefully inspected to ensure that all steps have been satisfactorily performed until then. After this initial phase of the surgical procedure, the defects will be randomized. For the GAP + OFD/EMD and GCP + OFD/EMD groups, there will be the application of EMD in the defect. For this, the surface in question should be free of saliva and blood. This substance will be applied immediately to the exposed root surface. The application will begin at the most apical portion of the bone level until the total coverage of the defect and the root surface. The flaps will then be repositioned and sutured passively until the primary closure of the tissues.

   Postoperative care: Patients will be instructed to take analgesic (sodium dipyrone 500mg every 4 hours for 2 days) and chelate 0.12% chlorhexidine digluconate (2 times a day for 15 days). The sutures will be removed after 15 days after the surgical procedure. During the postoperative period, the patient will be asked to stop brushing and flossing in the procedure area for 15 days, when the oral hygiene habits will be resumed.
7. Clinical evaluation

   The pre-calibration of the examiner for the measurements will be performed to ensure the reliability of the data obtained through two exams, with a maximum interval of 48 hours between them, in 8 different non-research patients. Kappa index and intraclass correlation will be used to evaluate reproducibility and agreement.

   All clinical parameters will be obtained using a North Carolina-type periodontal probe, at baseline, 3, 6 months and 1 year thereafter, with the aid of stents/individual acrylic guides, made from preformed study models by the examiner.

   The clinical parameters evaluated will be: Plate Index - PI; Bleeding on probing - BoP; Gingival margin position - GMP: distance from the stent to the free gingival margin; Relative Clinical Attachement Leval - rCAL: distance from the stent to the clinically detectable base of the periodontal pocket; Probing Depth - PD (rCAL - GMP): distance from the gingival margin to the clinically detectable base of the periodontal pocket.

   At the trans-surgical time, the following measurements will be performed: Distance between the stent margin and the alveolar bone crest (BC-ST); Distance between the alveolar bone crest and the base of the defect (BC-BD), characterizing the vertical component of the intrabony defect; Distance from the alveolar bone crest to the root surface (BC-RS), characterizing the horizontal component of the defect.
8. Patient satisfaction and perception of therapy

   For the assessment of the patient's perception of the procedure performed and the postoperative period, they will receive a questionnaire 15 days after the procedure. The extent of discomfort and/or pain experienced during the transoperative period will be evaluated using a 100mm horizontal analogue visual scale (VAS), ranging from absence to extreme. Patients will also be instructed to quantify the amount of analgesic used. In addition, the extent of discomfort, radicular hypersensitivity, edema, hematoma, fever and interference with daily activities during the first postoperative week will be assessed in the same way. After 6 months of the surgical procedure, another questionnaire will be delivered to determine the individuals' perception regarding the results and the level of satisfaction with the treatment. The questionnaire will use a simplified scale to record treatment satisfaction in terms of aesthetic appearance of the treated tooth by selecting one of the following: Very satisfied, neutral, moderately satisfied, or dissatisfied. In addition, patients will be questioned about their perceptions regarding the results of therapy applied to the teeth in question, in terms of improvement in gingival bleeding, redness, edema and hygiene pattern. These parameters will also be evaluated through the VAS scale, 0 being no improvement and 100 being the maximum improvement. Oral Health Impact Profile-14 (OHIP-14) will also be used in order to have access to oral health-related quality of life, applied in pre-surgery and 6 months later. The dimensions of the impact are: functional limitation, physical pain, psychological discomfort, physical incapacity, psychological incapacity and disability to perform daily activities. An adaptation of the Post-Surgical Patient Satisfaction Questionnaire (PSPSQ) will also be applied to evaluate the patient's satisfaction with the surgical procedure in the postoperative period of 15 days and 6 months. This 3-item scale, with a response from 0 to 10 (0 = not at 10 = totally), is capable of evaluating the patient's short- and long-term satisfaction in the postoperative period.
9. Radiographic evaluation[

   Periapical radiographs of all intrabony defects will be performed at the baseline, after 6 months and 1 year, using the parallelism technique, by the same examiner. For the standardization of the images will be made occlusal records in chemically activated acrylic resin with radiographic positioners. A standard orthodontic wire of known size will be placed on the occlusal support at a specific position, and the image of this wire will be obtained on radiographs for correction of vertical and horizontal angulation during the analyzes.

   The X-rays will be performed by a digital system using flexible and reusable phosphor storage plates (PSP; 31mm x 41mm). The selection of the exposure time will occur according to the tooth related to the defect, since the apparatus to be used (Sommo X-ray of mobile column, tube: 70 kV, 7 mA, focal length: 20 cm, specifications: 800-1200 VA, 50-60 Hz; has a semi-automatic tooth selection system, with established exposure times ranging from 0.32 to 0.40 seconds. For reading the images will be used a specific scanner. The images obtained will then be stored in a computer until the moment of analysis. The default resolution will be 96x96 dpi and 32 bit. All images will be recorded in TIFF (.tif) format. Radiographic measurements of defects will be performed using specific software for image analysis. The radiographic angles of the defects will be evaluated and defined by two lines representing the root surface and the surface of the bone defect.

   The following linear radiographic parameters will be measured: cement-enamel junction distance (CEJ) to the base of the defect (BD) (CEJ-BD); Distance from the CEJ and the more coronal portion of the alveolar bone crest (BC) (CEJ-BC); Distance between BD and BC (BD-BC). Differences between the values found at 6 months and 1 year postoperatively and the baseline for CEJ-BD will indicate the amount of hard tissue filling of the infra-osseous defect. Differences between CEJ-BC and BD-BC will identify the amount of resorption of the bone crest and the depth of the intrabony defect, respectively
10. Microbiological evaluation

    The microbiological evaluation will be done through the polymerase chain reaction (PCR) of the real time type. This test will allow the quantitative detection of the following bacteria: P. gingivalis, T. forsythia, A. actinomycetemcomitans, P. micro and P. intermedia.

    Subgingival biofilm samples will be performed at the baseline, 3, 6 months and 1 year after the surgical procedure, by the same examiner. To do this, the teeth and faces previously selected for the surgical phase will be used. The area will be properly insulated with sterilized cotton rolls. The supragingival portion of the biofilm will be removed, and then samples of the subgingival biofilm will be obtained by placing sterile absorbent paper cones inside the pocket. After 30 seconds the paper cones will be removed and placed in micro-centrifuge tubes with Tris-EDTA solution, coded for each patient. The eppendorfs shall be maintained at -20 ° C until the test is performed.

    For DNA extraction, the microtubes will be vortexed and the paper cones removed with clinical clamp aid. Samples will be centrifuged for removal of the supernatant. 700 µL extraction buffer is added, further shaken and placed in a water bath for 30 minutes at 65 ° C. The next step will be to add 650 μl CIA, homogenize to an emulsion (20 times) and centrifuge at 12,000-15,000 rpm for 7 minutes. The aqueous phase will be transferred to a new 1.5 mL microtube, to which 200 µL of extraction buffer without proteinase K will be added. Homogenization will then be done for addition of 650 µL CIA. Further homogenization and centrifugation at 12,000-15,000 rpm is continued for 7 minutes. The aqueous phase will be transferred to a new tube, to which 650 μl CIA will be added, followed by centrifugation at 12,000-15,000 rpm for 7 minutes (repeat two more times if needed). The DNA will be precipitated with 1 volume of isopropanol at room temperature, then homogenized (20 times) and centrifuged at 12,000-15,000 rpm for 7 minutes. The surface of the precipitate will be washed once with 50 μl of 70% ethanol prepared shortly before use and then centrifuged for 2 minutes. The precipitate should be dried, leaving the tube open on bench next to Busen's nozzle. Afterwards, resuspension will be done in 40 μL TE (10 mM Tris-HCl, pH 8.0, 1 mM EDTA, pH 8.0) + 10 μg / mL RNAse and to leave in a water bath at 37 ° C for 30 minutes. Five μL of the sample will be used to check the quality and estimate the amount of DNA in a 0.8-1.0% agarose gel. A known mass standard (pGEM) will run together.

    Real time PCR DRAWING OF PRIMERS: Specific primers for Porphyromonas gingivalis, Tannerella forsythia, Parvimonas micra, Prevotella intermedia and A. actinomycetemcomitans will be used. All primers will be checked for specificity by checking the Melting curve (obtained after running in the LightCycler) and running gel for product verification.

    OPTIMIZATION OF REACTIONS: The use of SYBR Green I requires specific PCR products, so that the effectiveness of the primer reactions will be optimized prior to the initiation of the reactions themselves. Concentrations ranging from 2 to 5 mM MgCl2 and from 0.2 to 0.5 μM of each primer will be used to determine under what conditions the reaction would have the best efficiency. Conditions suggested by the equipment manufacturer.

    RT-PCR reactions: RT-PCR reactions will be performed with the LightCycler system using the FastStart DNA Master SYBR Green I kit. The reaction profile will be determined following the equipment manufacturer's recommendations. For each of the "runs", the water will be used as a negative control, and the reaction product will be quantified using the manufacturer's own program.
11. Immunoenzymatic test (Luminex platform / MAGpix)

    Gingival Crevicular Fluid (GCF) collections will be performed at the baseline, 15, 45 days, 3, 6 months and 1 year after the study, by the same examiner. To do this, the teeth and faces previously selected for the surgical phase will be used. During collection of the material, the site involved will be properly insulated and dried with sterilized cotton rolls. The supragingival portion of the bacterial biofilm will be removed to obtain GCF samples by placing paper strips within the tooth / periodontal tissue interface for 30 seconds. Two strips of paper per site will be used for obtaining suitable and the paper strips will then be placed in microcentrifuge tubes, coded for each individual and experimental periods with 150 μl of phosphate buffered saline (PBS) and 0.05% Tween-20. The samples will be stored for further analysis.

    Prior to analysis, the fluid samples will be diluted in 60μl of buffer from the Millipore kit, vortexed for 30 minutes and then centrifuged for 10 minutes at 10,000 rpm. Aliquots of each GCF sample will be analyzed for the detection of bone markers (PDGF, VEGF, FGF, OPG, OCN, OPN, TGFα, PTH and RANKL) by Luminex / MAGpix technology. To do so, the analyzes will be performed in 96 well plates with the aid of high sensitivity panels, following the manufacturer's instructions. Briefly, the wells will be washed with wash buffer and aspirated. Exclusive microspheres conjugated to monoclonal antibodies against the different analytes to be analyzed will be added to the wells (the polystyrene microspheres are stained with precise proportions of two fluorophores, creating a "color code" for further identification by the Luminex / MAGpix instrument). Samples and reagents for the standard curve will be pipetted into the wells and incubated overnight at 4oC. The wells will then be washed and a mixture of secondary antibodies will be added. After incubation for 1 hour, the final detection will be done through a third fluorescent label, Streptavidin-Phycoerythrin (PE) bound to the detection antibody. The Luminex / MAGpix equipment will move these beads in single file through bundles of two different lasers on a flow cytometer. The first laser beam will detect (classify) the microsphere (the color code for the test) and the second laser will quantify the reporting signal in each microsphere. Samples will be individually analyzed and their concentrations will be estimated from a standard curve using a polynomial equation using Xponent software. The mean concentrations of each marker will be expressed in pg / μl. Samples with quantification below the detection limit of the analysis shall be recorded as "zero" and samples above the limit of quantification of the standard curve shall be recorded equal to the highest value of the curve.
12. Analysis of results The analysis of the results will be done through descriptive statistics using tables and graphs containing absolute and relative frequencies and parameters of mean and standard deviation. The comparison of the quantitative variables will be done through analysis of variance and Tukey's test. Qualitative variables will be compared using the chi-square test. The correlation check between the variables will be done through the Pearson and Spearman correlation coefficient. In all tests, a significance level of 5% will be adopted.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of generalized aggressive periodontitis (verified by the presence of periodontal pockets and radiological loss in patients under the 35 years old at the time of diagnosis); or a diagnosis of generalized chronic periodontitis (in patients over 35 years old);
* Presence of infra-osseous defect in radiographic examination with minimum dimensions of 4mm deep and 2mm of horizontal component, associated to periodontal pocket of at least 6mm of PD;
* Presence of at least 15 teeth of the oral cavity;
* To present less than 20% of plaque index and bleeding on probing after 6 weeks of initial therapy;
* Formal consent for participation in research, after explaining the risks and benefits for individual not involved in it. (Resolution No. 196 of October 1996 and the Dental Code of Professional Ethics (C.F.O.) 179/93).

Exclusion Criteria:

Presence of periapical or pulpal alteration;

* Presence of systemic alteration or use of medications (6 months prior to the study) that may influence the response to periodontal treatment;
* Pregnant and lactating women;
* Smoking;
* Periodontal treatment including subgingival instrumentation in the 6 weeks prior to the study;
* Teeth with bifurcation involvement;
* Teeth with marked mobility;
* Oral pathology, chronic disease or history of allergy to any component of the study;
* Previous periodontal surgery in the region of interest.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Relative Clinical Attachment Level | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ana Lívia F Santana, MD, Principal Investigator — School of Odontology of Piracicaba - Unicamp
Locations (1):
- Piracicaba Dental School, State University of Campinas, Piracicaba, São Paulo, Brazil